CLINICAL TRIAL: NCT04217356
Title: A Patient Preferences-Controlled Study of Allogeneic Hematopoietic Cell Transplantation Versus Best Available Non-Transplant Therapies in Patients With High-Risk Myelofibrosis (ALLO-BAT Study)
Brief Title: Study of Stem Cell Transplant vs. Non-Transplant Therapies in High-Risk Myelofibrosis
Acronym: ALLO-BAT
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 19-6362; ALLO-BAT (Other: Princess Margaret Cancer Centre)
Record Dates: First submitted 2020-01-02; First posted 2020-01-03 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Myelofibrosis; High-Risk Cancer; Bone Marrow Cancer
Keywords: High-Risk Myelofibrosis; Stem Cell; Transplantation; Myelofibrosis; Bone marrow cancer
MeSH Terms: conditions — Primary Myelofibrosis; Bone Marrow Neoplasms | interventions — Stem Cell Transplantation; ruxolitinib; Hydroxyurea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for future research related to hematological (blood) cancers and their treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hematopoietic stem cell transplant (HCT): Standard of care hematopoietic stem cell transplant with a matched donor.
  Interventions: Biological: Hematopoietic stem cell transplant
- Best available non-transplant therapies (BAT): Standard of care treatment with a janus kinase (JAK) inhibitor drug called ruxolitinib or treatment with an antimetabolite drug called hydroxyurea.
  Interventions: Drug: Ruxolitinib; Drug: Hydroxyurea

INTERVENTIONS:
Biological: Hematopoietic stem cell transplant — Intravenous infusion of hematopoietic stem cells from a donor.
  Groups: Hematopoietic stem cell transplant (HCT)
Drug: Ruxolitinib — Ruxolitinib is type of drug called a janus kinase (JAK) inhibitor. Ruxolitinib is taken orally (by mouth).
  Other Names: JAKAVI
  Groups: Best available non-transplant therapies (BAT)
Drug: Hydroxyurea — Hydroxyurea is a type of drug called an antimetabolite. Hydroxyurea is taken orally (by mouth).
  Groups: Best available non-transplant therapies (BAT)

SUMMARY:
The purpose of this research study is to see how effective hematopoietic stem cell transplantation (HCT) is compared to best available non-transplant therapies (BAT) in patients with high risk myelofibrosis. This will be done by asking participants to choose the treatment that they prefer to receive (HCT or BAT) and then comparing the outcomes of the participants in both treatment groups.

DETAILED DESCRIPTION:
There is currently little information regarding which treatments are best for patients with myelofibrosis. On one hand, hematopoietic stem cell transplantation (HCT) is potentially curative treatment but is associated with significant risk of complications related to graft failure (the new donor cells does not grow properly after the transplant), side effects such as graft versus host disease (the patient's cells attack the new donor cells), and risk of infections. Non-transplant therapies such as ruxolitinib provide effective symptom control for few months to few years, but are not curative in nature. As such, this study will compare the effectiveness of HCT versus best available non-transplant therapies (BAT) in patients with high risk myelofibrosis.

This is an observational study, meaning that participants will be followed to assess the effects of their treatment, but no intervention (treatments) will be given as a part of this study.

ELIGIBILITY:
Inclusion Criteria:

Recruitment Part:

* Documented diagnosis of pre-fibrotic primary myelofibrosis (pre-fibrotic PMF), overt PMF, post-polycythemia MF (PPV-MF) or post-essential thrombocythemia MF (PET-MF) confirmed by bone marrow biopsy
* Have been tested or have results available for phenotypic driver mutations (JAK2/CALR/MPL) and high molecular risk (HMR) mutations using a broad myeloid malignancies targeted gene panel.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Able to provide informed consent
* Adequate organ function
* Donor search initiated or patient is agreeable to donor search
* Meet the definition/criteria for high-risk myelofibrosis

Study Arm Allocation:

* Grade of fibrosis on bone marrow biopsy available according to World Health Organization (WHO) criteria
* Results available for phenotypic driver mutations (JAK2/CALR/MPL) and targeted sequencing results using a broad myeloid malignancy panel with a minimal requirement to include results on High molecular risk (HMR) mutations such as ASXL1/EZH2/IDH1/IDH2/SRSF2/U2AF1/TP53
* ECOG performance status 0-2
* Adequate organ function
* Information on donor search and donor type available

Exclusion Criteria:

Recruitment Part:

* Blasts in peripheral blood or bone marrow ≥10%
* For patients already on ruxolitinib at study entry, and meet the criteria of ruxolitinib failure
* Previous history of transformation to blast phase or acute myeloid leukemia
* Received allogeneic stem cell transplant for myeloproliferative neoplasm
* Presence of an active uncontrolled infection
* Myocardial infarction in the preceding 3 months
* Active hepatitis A, B or C
* Known human immunodeficiency virus (HIV) positive
* History of active malignancy in the previous 2 years, except basal cell carcinoma or squamous cell carcinoma of skin or stage 0 cervical cancer
* Any psychiatric illness or social circumstances or significant co-morbid conditions that will prevent patient from proceeding to allogeneic hematopoietic cell transplantation.
* Pregnant or breastfeeding women

Study Arm Allocation:

* Blasts in peripheral blood or bone marrow ≥10%
* Meet the criteria of ruxolitinib failure
* Presence of an active uncontrolled infection
* Myocardial infarction in the preceding 3 months
* Active hepatitis A, B or C
* Known HIV positive
* History of active malignancy in the previous 2 years, except basal cell carcinoma or squamous cell carcinoma of skin or stage 0 cervical cancer
* Pregnant or breastfeeding women
* Any psychiatric illness or social circumstances or significant co-morbid conditions that will prevent patient from proceeding to allogeneic hematopoietic cell transplantation.
* Time between registration and allocation of study arm >24 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high-risk myelofibrosis including pre-fibrotic primary myelofibrosis (pre-fibrotic primary myelofibrosis), overt primary myelofibrosis, post-polycythemia myelofibrosis or post-essential thrombocythemia myelofibrosis.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-08-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients allocated to hematopoietic stem cell transplantation (HCT) | 5 years
Number of patients allocated to best available non-transplant therapies (BAT) | 5 years
Overall survival rate of patients who receive hematopoietic stem cell transplantation (HCT) | 5 years
  Time from study allocation to death or last follow up.
Overall survival rate of patients who receive best available non-transplant therapies (BAT) | 5 years
  Time from study allocation to death or last follow up.

SECONDARY OUTCOMES:
Median change in Patient Global Impression of Change (PGIC) score | 0 and 36 months
  Range from -3 to 3. Positive number equals increase in quality of life.
Median change in MPN Symptom Assessment Form Total Symptom Score (MPN-SAF TSS) | 0 and 36 months
  Range from 0 to 10. Increase equals worsening of symptoms.
Median change in FACT-BMT Questionnaire | 0 and 36 months
  Range from 1 to 4. Increase equals increase in quality of life.
Disease-free survival of patients who receive hematopoietic stem cell transplantation (HCT) | 5 years
  Time from allocation to study arm to death/acute myeloid leukemia transformation or last follow up.
Disease-free survival of patients who receive best available non-transplant therapies (BAT) | 5 years
  Time from allocation to study arm to death/acute myeloid leukemia transformation or last follow up.
Number of patients who receive hematopoietic stem cell transplantation (HCT) in remission (complete and partial) | 3 years
Number of patients who receive best available non-transplant therapies (BAT) in remission (complete and partial) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Gupta, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (5):
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No